CLINICAL TRIAL: NCT07320391
Title: Comparison of Topically Applied Ozonated Gel and Titanium Platelet-rich Fibrin (Tprf) on Palatal Wound Healing (A Randomized Controlled Clinical Trial)
Brief Title: Ozonated Gel and Titanium Platelet-rich Fibrin (on Palatal Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0968_ 09/2024
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Palatal Lesion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ozonated gel (Experimental)
  Interventions: Other: Ozonated Gel Application
- Application of TPRF (Active Comparator)
  Interventions: Other: T-PRF Application
- flowable composite (Other)
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Ozonated Gel Application — After harvesting the free palatal grafts, an adrenaline-soaked sterile surgical gauze was applied to the palatal donor sites with firm pressure for 5 minutes to achieve hemostasis. Subsequently, ozonated gel loaded on gelatin foam was placed over the donor sites and stabilized using flowable composite.
  Arms: ozonated gel
Other: T-PRF Application — Twenty milliliters of venous blood were collected from the antecubital vein and immediately centrifuged at 2800 rpm for 12 minutes. The resulting T-PRF clots were retrieved using sterile tweezers, separated from the red blood cell layer, and placed on sterile woven gauze. The clots were allowed to exude serum for 20 minutes, then gently compressed between gauze to form T-PRF membranes. The membranes were trimmed to fit the FGG donor site and covered with flowable composite.
  Arms: Application of TPRF
Other: Conventional treatment — After harvesting the free palatal grafts, an adrenaline-soaked sterile surgical gauze was applied to the palatal wounds with firm pressure for 5 minutes to achieve hemostasis. The palatal wounds were then covered with flowable composite.
  Arms: flowable composite

SUMMARY:
Background: autogenous soft tissue grafts can be considered the gold standard for treatment of mucogingival problems. The most common site for harvesting the graft is the palate. The palatal donor site for free gingival graft (FGG) significantly influences the pain and discomfort experienced by the patient, and there is a potential for postoperative bleeding.To overcome these problems many dressing materials associated with topical formulae have been used.

Aim: The objective of this study is to assess the effect of topically applied ozonated oil on palatal wound healing and compare it to the effect of titanium platelet rich fibrin (TPRF)

ELIGIBILITY:
Inclusion Criteria:

* Isolated gingival recession defects on the mandibular and maxillary anterior teeth with insufficient keratinized gingiva.
* Good oral hygiene

Exclusion Criteria:

* Patients reporting systemic conditions that may compromise healing or bone metabolism
* Patients having a history of radiotherapy, chemotherapy or bisphosphonate therapy.
* Pregnant women or those planning to get pregnant during the study course
* History of periodontal disease or previous periodontal surgery on the experimental sites
* Smoking or any other deleterious habits.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in pain scores | Up to 14 days
  Patients will be asked to grade the severity of pain using VAS. It ranges across a continuum from none to an extreme amount of pain in a straight horizontal 10 cm line [from 0-100 mm].
Change in wound area | Baseline, 3 days, 7 days, 10 days, and 14 days
  Standardized clinical photographs of the palatal surgical sites will be obtained on the day of surgery and at 3, 7, 10, and 14 days postoperatively. Photographs will be taken perpendicular to the wound area, with a standard-sized visual scale placed adjacent to the palatal wounds to allow accurate wound size measurement and analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Periodontology and Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt